CLINICAL TRIAL: NCT06036485
Title: Efficacy of Kerecis Omega 3 Versus Standard of Care in Patients With Chronic Leg Ulcerations - a Randomized Trial With a New In-wound Split Design Approach
Brief Title: Efficacy of Kerecis Omega 3 in Comparison to Clinical Standard Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to support the study
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kerecis-1
Record Dates: First submitted 2023-03-15; First posted 2023-09-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Intervention Model Description: 1:1 in-wound split design with random allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kerecis Omega 3 (Experimental)
  Interventions: Device: Kerecis Omega 3
- Surgical debridement (Active Comparator)
  Interventions: Procedure: Surgical debridement

INTERVENTIONS:
Device: Kerecis Omega 3 — Decellularized intact fish skin developed for the management of chronic wounds
  Arms: Kerecis Omega 3
Procedure: Surgical debridement — Superficial sharp surgical debridement technique
  Arms: Surgical debridement

SUMMARY:
Chronic leg ulcerations are a great burden for patients and the medical system alike. Frequent outpatient consultations with associated treatment costs and travel costs for the patient as well as psychosocial burdens remain an unmet problem in chronic wound care. There is an increasing need for definitive treatment of especially chronic venous and multifactorial chronic leg ulceration where arterial intervention is not a treatment option.

Minimal invasive surgical interventions that do not require skin grafting can be performed under local anesthesia in an outpatient setting even in multimorbid patients.

Kerecis Omega3 Wound is intact decellularized fish skin. The fish skin sheets contain fat, protein, elastin, glycans and other natural skin elements and it can be an effective treatment option in chronic leg ulcerations and is licensed for this use as a medical product in Switzerland. However, limited data without inter-wound bias is available for the use of Kerecis Omega 3 in chronic leg ulcerations.

In this study the investigators propose to investigate the efficacy of Kerecis Omega 3 according to objective wound surface measurements using standardized digital photographs in patients with chronic leg ulcerations. Efficacy will be evaluated against standard of care wound debridement.

ELIGIBILITY:
Inclusion Criteria:

* Any chronic leg ulcer > 4 weeks duration with delayed wound healing (reduction of wound surface of less than 40-50% within 4 weeks under adequate local therapy) without underlying treatable medical conditions
* Ulcer area at between 5cm2 and 60cm2
* Bacterial swab sampling prior to study
* Written study informed consent

Exclusion Criteria:

* History of Fish allergy or proven Fish allergy
* Pregnant or breast-feeding women
* Intention to become pregnant during the course of the study
* Wound not suitable for dressing: inflammation, fibrin coatings
* Inability to understand the study consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in ulcer surface area | 12 weeks
  Change in ulcer surface area as assessed by standardized photography and digital imaging.

SECONDARY OUTCOMES:
Change in patient quality of life | 2, 4, 6 and 12 weeks
  Change in patient quality of life as assessed by the Wound-QoL questionnaire score, ranging from 0 to 4, with higher scores indicating a worse quality of life.
Change in wound microbiota as assessed by alpha diversity of the microbial composition | 2, 4, 6 and 12 weeks
  Change in wound microbiota utilizing 16S-sequencing from wound swabs as assessed by alpha diversity of the microbial composition trough Shannon index, with higher scores indicating a more diversity of the species
Change in wound microbiota as assessed by beta diversity of the microbial composition | 2, 4, 6 and 12 weeks
  Change in wound microbiota utilizing 16S-sequencing from wound swabs as assessed by beta diversity of the microbial composition trough Shannon index, with higher scores indicating a more diversity of the species.
Change in ulcer surface area | 2, 4, 6 and 12 weeks
  Change in ulcer surface area as assessed by standardized photography and digital imaging.

OTHER OUTCOMES:
Incidence of adverse events | 12 weeks
  Cumulative incidence of treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bossart, MD, Principal Investigator — Department of dermatology, University Hospital Inselspital, Bern

IPD SHARING:
Plan to Share IPD: No